CLINICAL TRIAL: NCT01697306
Title: The Impact of Intravesical Gemcitabine and 1/3 Dose Bacillus-Calmette Guerin (BCG) Instillation Therapy on the Quality of Life in Non-muscle-invasive Bladder Cancer (NMIBC) Patients: Results of a Prospective, Randomised Phase II Trial.
Brief Title: The Impact of Intravesical Gemcitabine and 1/3 Dose Bacillus Calmette-Guerin on the Quality of Life in Superficial Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: University of Turin, Italy (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Marco Oderda, MD, Azienda Ospedaliera San Giovanni Battista
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CE 70/06
Record Dates: First submitted 2012-09-21; First posted 2012-10-02 (Estimated); Last update posted 2025-01-30 (Actual); Status verified 2012-09

CONDITIONS: Bladder Cancer
Keywords: non muscle invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine; BCG Vaccine; BCG Connaught

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine-arm (Active Comparator): 7-15 days after TUR patients received six weekly instillations of gemcitabine (Gemzar, Eli Lilly SpA), 2.000 mg diluted in 50 cc of saline. Maintenance consisted in monthly instillations up to 1 year
  Interventions: Drug: Gemcitabine 2 g
- BCG-arm (Active Comparator): 7-15 days after TUR patients received an induction cycle of six weekly instillations of Connaught strain Bacillus Calmette-Guerin (BCG Immucyst) 1/3 dose (27 mg) diluted in 50 cc of saline. Maintenance consisted of 3 weekly instillations at 3, 6 and 12 months
  Interventions: Drug: BCG Vaccine

INTERVENTIONS:
Drug: Gemcitabine 2 g — six weekly instillations of gemcitabine (Gemzar, Eli Lilly SpA), 2.000 mg diluted in 50 cc of saline
  Other Names: Gemzar, Eli Lilly SpA
  Arms: Gemcitabine-arm
Drug: BCG Vaccine — six weekly instillations of Connaught strain BCG (Immucyst) 1/3 dose (27 mg) diluted in 50 cc of saline
  Other Names: BCG Connaught 1/3 dose
  Arms: BCG-arm

SUMMARY:
To our knowledge, there are no comparative studies on bacillus Calmette-Guerin (BCG) and intravesical chemotherapy addressing quality of life (QoL) issues. The aim of this study was to prospectively evaluate and compare the QoL of intermediate-risk non-muscle-invasive (NMIBC) patients treated with BCG or gemcitabine.

DETAILED DESCRIPTION:
Intravesical Bacillus Calmette-Guérin (BCG) is considered the most effective agent for non-muscle-invasive bladder cancer (NMIBC), representing the first-line option in the management of carcinoma in situ (CIS) and high-risk disease. In intermediate-risk NMIBC, however, both BCG and intravesical chemotherapy are accepted alternative adjuvant options since the superiority of BCG has been only established for disease recurrence but not progression and it needs to be balanced against higher toxicity. According to current evidence, BCG is considered less tolerable than intravesical chemotherapy such as mitomycin-C or doxorubicin, based on reported side effects. Among chemotherapeutic agents, gemcitabine has an excellent toxicity profile and promising efficacy in NMIBC patients, including those at high-risk of disease recurrence, even if its role on the management of NMIBC has not been well-defined yet. To our knowledge, there are no comparative studies on BCG and intravesical chemotherapy addressing quality of life (QoL) issues. The aim of this study was to prospectively evaluate and compare the QoL of intermediate-risk NMIBC patients treated with BCG or gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical evidence of intermediate-risk non-muscle invasive bladder cancer (namely Ta-1, G1-2, multifocal or unique and recurrent, >3 cm in diameter)
* WHO performance status ≤2
* age ≤85years
* BCG naive
* patients not treated with intravesical chemotherapy in the last 3 months.

Exclusion Criteria:

* presence of T1G3 or CIS
* preoperative urinary cytology positive for high-grade atypia
* inadequate bone marrow reserve (white blood cells <3 x 109/l, platelets <100 x 109/l)
* history of genito-urinary tuberculosis
* presence of uncontrolled urinary infections.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-09; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
quality of life of intermediate-risk NMIBC patients treated with intravesical Gemcitabine chemotherapy or BCG | 1 year

SECONDARY OUTCOMES:
comparison of the short term efficacy of the two treatments in terms of recurrence | 1 year
comparison of the short term efficacy of the two treatments in terms of progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Gontero, Professor, Principal Investigator — A.O.U. San Giovanni Battista Molinette
Locations (1):
- A.O.U. San Giovanni Battista Molinette, Torino, TO, Italy

REFERENCES:
- [Background] Martinez-Pineiro JA, Martinez-Pineiro L, Solsona E, Rodriguez RH, Gomez JM, Martin MG, Molina JR, Collado AG, Flores N, Isorna S, Pertusa C, Rabadan M, Astobieta A, Camacho JE, Arribas S, Madero R; Club Urologico Espanol de Tratamiento Oncologico (CUETO). Has a 3-fold decreased dose of bacillus Calmette-Guerin the same efficacy against recurrences and progression of T1G3 and Tis bladder tumors than the standard dose? Results of a prospective randomized trial. J Urol. 2005 Oct;174(4 Pt 1):1242-7. doi: 10.1097/01.ju.0000173919.28835.aa. PMID 16145378
- [Background] Porena M, Del Zingaro M, Lazzeri M, Mearini L, Giannantoni A, Bini V, Costantini E. Bacillus Calmette-Guerin versus gemcitabine for intravesical therapy in high-risk superficial bladder cancer: a randomised prospective study. Urol Int. 2010;84(1):23-7. doi: 10.1159/000273461. Epub 2010 Feb 17. PMID 20173364